CLINICAL TRIAL: NCT03629080
Title: A Randomized, Placebo-Controlled, Phase 2 Study of HB-101, a Bivalent Cytomegalovirus (CMV) Vaccine, in CMV-Seronegative Recipient (R-) Patients Awaiting Kidney Transplantation From Living CMV-Seropositive Donors (D+).
Brief Title: A Study of CMV Vaccine (HB-101) in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-100-002; 2017-005047-32 (EudraCT Number)
Record Dates: First submitted 2018-05-29; First posted 2018-08-14 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cytomegalovirus (CMV) Infection; Kidney Transplantation
Keywords: solid organ transplantation; vaccine
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: This phase 2 study will be conducted in three groups stratified by treatment intent. In Group 1, patients will be randomized to receive HB-101 (1a) or placebo (1b) and followed preemptively post-transplant. Approximately 50 patients will be randomized in Group 1. In Group 2, patients will be randomized to receive HB-101 (2a) or placebo (2b) before transplant. Post-transplant patients will receive 3-6 months of anti-viral prophylaxis following institutional standards. Approximately 100 patients will be randomized in Group 2. In Group 3, all patients will receive HB-101 (open label) vaccination(s) prior to their transplant surgery. Post-transplant CMV management will follow either preemptive or prophylactic care as defined at study enrollment by the investigator and institutional standards. Approximately 25 patients will be randomized in Group 3.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants, investigators and care providers (study site personnel) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- HB-101 vaccine preemptive (Experimental): Three doses of HB-101 vaccine will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of HB-101 will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post-transplant patients will be monitored per preemptive institutional standard.
  Interventions: Biological: HB-101 vaccine
- Placebo preemptive (Placebo Comparator): Three doses of placebo will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of placebo will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post-transplant patients will be monitored per preemptive institutional standard.
  Interventions: Biological: placebo
- HB-101 vaccine prophylactic (Experimental): Three doses of HB-101 will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of HB-101 will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post- transplant patients will receive 3-6 months anti-viral prophylaxis following institutional standard.
  Interventions: Biological: HB-101 vaccine
- Placebo prophylactic (Placebo Comparator): Three doses of placebo will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of placebo will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post- transplant patients will receive 3-6 months anti-viral prophylaxis following institutional standard.
  Interventions: Biological: placebo
- HB-101 vaccine: CMV (+) patients-Prophylactic Management (Experimental): Three doses of HB-101 will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of HB-101 will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post- transplant patients will receive 3-6 months anti-viral prophylaxis following institutional standard.
  Interventions: Biological: HB-101 vaccine
- HB-101 vaccine: CMV (+) patients-Preemptive Management (Experimental): Three doses of HB-101 will be administered prior to transplantation and within proximity to the time of transplantation. However, two doses of HB-101 will be sufficient for the patients to be included in the efficacy analyses if an administration of the third dose is not feasible due to transplantation timelines. Post- transplant patients will follow pre-emptive management per institutional standard.
  Interventions: Biological: HB-101 vaccine

INTERVENTIONS:
Biological: HB-101 vaccine — HB-101 is a bivalent vaccine that contains two replication deficient recombinant lymphocytic choriomeningitis virus (rLCMV) vectors expressing pp65 and a truncated isoform of gB of human CMV.
  Arms: HB-101 vaccine preemptive; HB-101 vaccine prophylactic; HB-101 vaccine: CMV (+) patients-Preemptive Management; HB-101 vaccine: CMV (+) patients-Prophylactic Management
Biological: placebo — Saline will be used for placebo.
  Arms: Placebo preemptive; Placebo prophylactic

SUMMARY:
HB-101 is a bivalent recombinant vaccine against human CMV infection. This is a randomized, placebo-controlled, phase 2 study to assess the safety, reactogenicity, immunogenicity, and efficacy of HB-101 in CMV-Seronegative patients receiving a kidney transplant from a CMV-Seropositive living donor and CMV-Seropositive patients.Patients enrolled should have a living donor kidney transplantation ideally planned between two to four months after the first injection of study drug (HB-101 or placebo).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, phase 2 study to assess the safety, reactogenicity, immunogenicity, and efficacy of HB-101 in adult patients awaiting kidney transplantation. For Groups 1 and 2, adult CMV-seronegative (-) patients awaiting kidney transplant from a CMV-seropositive (+) living donor will be enrolled according to treatment intent with regard to the method of CMV prevention after transplant (either preemptive or prophylactic). This will be defined at study enrollment by the investigator and institutional standards. Patients enrolled in Group 1 and 2 will be randomized to receive HB-101 or placebo. For Group 3, adult CMV-seropositive (+) patients awaiting kidney transplant from either CMV-seropositive(+) or CMV-seronegative(-) living donors will be enrolled. Group 3 will be open label where all patients will receive HB-101. The post transplant management for Group 3 patients will also follow either preemptive or prophylactic method per the institution standards. The intent of the study is to administer three doses of the study drug (HB-101 or placebo) prior to transplantation and within proximity to the time of transplantation. However, two doses of study drug will be sufficient for the patients to be included in the efficacy analyses if a third dose of study drug is not feasible due to transplantation timelines. Patients will not receive study drug after transplantation. Patients will be recruited globally from transplant centers. The total duration of the study of each patient participating in the study will be approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following key inclusion criteria will be eligible to participate in the study:

1. Male or female patients 18 years of age or older.
2. Patients must be eligible to undergo kidney transplantation from a living donor as per institutional standards.
3. For Groups 1 and 2 only: Patients must be CMV immunoglobulin G (IgG) seronegative (-) and receiving kidney for transplantation from donors who are CMV IgG seropositive (+).
4. For Group 3 only: Patients must be CMV immunoglobulin G (IgG) seropositive (+) and receiving kidney for transplantation from donors who are either CMV IgG seronegative (-) or seropositive (+).
5. Patients who would comply with the requirements of this protocol (e.g., return for follow up visits), as judged by the investigator.

Exclusion Criteria:

Patients who meet any of the following key criteria will be excluded from the study:

1. Patients planning to undergo multi-organ transplantation.
2. Patients participating in another interventional clinical study.
3. Previous vaccination with an investigational CMV vaccine.
4. Any confirmed or suspected immunodeficiency disorder (based on medical history and physical examination) that could interfere with the immune response or that presents a risk for the patient to receive a vaccine candidate in development.
5. Treatment with any chronic immunosuppressive medication or other immuno modifying drugs within 6 months prior to study entry. However, inhaled and topical steroids and low-dose oral corticosteroids (<10 milligrams a day of prednisone or equivalent) are allowed.
6. Prior history of CMV disease or CMV infection requiring anti-viral therapy
7. Patients with a rash, dermatological condition, or tattoo in the area of the injection site(s) that could interfere with administration site reaction rating. (Note: The injection site(s) can be the non-dominant arm [most preferred injection site], dominant arm, or either thigh [least preferred injection site], as judged by the investigator).
8. It is anticipated that the patient will be unavailable to complete the study follow-up.
9. Patients who are highly sensitized or who are likely to undergo desensitization at time of transplant (e.g., donor-specific antibody titers at the local laboratory >2000).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Hookipa Biotech GmbH
Locations (25):
- United States (13):
  - The 1917 Clinic at UAB, Birmingham, Alabama
  - California Institute of Renal Research, La Mesa, California
  - UC Davis Health Systems, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Indiana University/IU Health, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati (UC) - College of Medicine, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - Thomas E. Starzl Transplantation Institute, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- Odense University Hospital, Odense, Denmark
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux Hôpital Pellegrin, Bordeaux
  - Hopital Necker-Enfants Malades, Paris
  - CHU de Toulouse - Hospital Rangueil, Toulouse
- Germany (2):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Essen, Essen
- Oslo University Hospital, Oslo, Norway
- United Kingdom (5):
  - Belfast Health and Social Care Trust, Belfast
  - Cardiff & Vale University Health Board, Cardiff
  - St James's University Hospital, Leeds
  - Leicester General Hospital, Leicester
  - The Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Started | 12 | 5 | 35 | 17 | 10 | 4
Completed | 10 | 4 | 22 | 16 | 6 | 3
Not Completed | 2 | 1 | 13 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management | Total
Number analyzed (Participants) | 12 | 5 | 35 | 17 | 10 | 4 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 31 | 16 | 9 | 4 | 71
  >=65 years | 3 | 3 | 4 | 1 | 1 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (15.9) | 63.6 (9.45) | 47.3 (15.13) | 45.5 (13.99) | 49.5 (11.92) | 48.3 (6.99) | 48.31 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 6 | 6 | 3 | 1 | 20
  Male | 8 | 5 | 29 | 11 | 7 | 3 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 4 | 0 | 1 | 0 | 10
  Not Hispanic or Latino | 12 | 0 | 29 | 16 | 6 | 2 | 65
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 3 | 0 | 0 | 0 | 3
  White | 11 | 5 | 28 | 17 | 8 | 4 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assess the number and severity of participants with adverse events and serious adverse events
Time Frame: 15 Months
Population: For the safety population: In groups "HB-101 prophylactic", "Placebo prophylactic" and "placebo preemptive" each 1 subject was excluded for reason being not receiving any study drug. One patient who was randomized to HB-101, received 2 doses of placebo and as a result, this patient was included in the placebo
Measure: Count of Participants; unit: Participants
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 11 | 4 | 34 | 17 | 10 | 4
Participants
  Adverse Events | 6 | 3 | 23 | 12 | 6 | 3
  Serious Adverse Events | 5 | 2 | 14 | 5 | 2 | 2
  Grade 3 or Higher Adverse Events | 0 | 0 | 0 | 0 | 2 | 2

2. Primary Outcome: Assessment of Humoral Immunogenicity Analyses
Description: Assessment of CMV neutralizing antibody titers (NTAs) at day of Transplant defined by log10 virus neutralising unit(s)
Time Frame: 15 Months
Population: The modified intent to treat population includes all participants who received a kidney transplant and at least 2 doses of study drug prior to kidney transplant.
Measure: Mean (Full Range); unit: log10 neutralizing titers
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
log10 neutralizing titers
  CMV Neut (2 Doses): number analyzed (Participants) | 6 | 2 | 15 | 7 | 4 | 1
  CMV Neut (2 Doses) | 0.8 [0.6 to 1.2] | 0.6 [0.6 to 0.6] | 0.8 [0.6 to 1.8] | 0.8 [0.6 to 1.7] | 2.6 [2.5 to 2.7] | 2.5 [2.5 to 2.5]
  CMV Neut (3 Doses): number analyzed (Participants) | 2 | 2 | 5 | 6 | 1 | 2
  CMV Neut (3 Doses) | 1.1 [0.6 to 1.5] | 0.6 [0.6 to 0.6] | 1.4 [1.2 to 1.8] | 0.6 [0.6 to 0.6] | 2.7 [2.7 to 2.7] | 2.5 [2.2 to 2.8]

3. Primary Outcome: Number of Patients With Injection Site Events.
Description: Number of patients experiencing a local or generalized injection site reaction
Time Frame: 15 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 11 | 4 | 34 | 17 | 10 | 4
Participants | 1 | 0 | 4 | 4 | 2 | 1

4. Primary Outcome: Change of Oral Body Temperature.
Description: Oral body temperature was measured in degrees Celsius prior to study drug administrations and seven days after. The results express the change from baseline (defined as the last measurement prior to the first dose of study drug) to Dose 3.
Time Frame: Change from Baseline to 7 days after study drug administration of Dose 3. Three (3) months
Population: Only participants having received all 3 doses are analyzed and presented.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 3 | 1 | 12 | 7 | 1 | 2
Degrees Celcius | -0.0 (0.4) | -0.1 (0.0) | 0.2 (0.6) | -0.3 (0.26) | 0.6 (0.0) | -0.2 (0.57)

5. Primary Outcome: Change of Respiration Rate.
Description: Respiration rate in breaths per minute was measured prior to study drug administration and seven days after. The results express the change from baseline (defined as the last measurement prior to the first dose of study drug) to Dose 3.
Time Frame: Change from Baseline to 7 days after study drug administration of Dose 3. Three (3) months.
Population: Only participants having received all 3 doses are analyzed and presented.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 4 | 1 | 11 | 7 | 1 | 2
breaths/minute | 0.5 (5.26) | 0.0 (0.0) | 0.2 (2.56) | -0.6 (2.70) | 2.0 (0.0) | -4.0 (8.49)

6. Primary Outcome: Change of Blood Pressure.
Description: Diastolic and Systolic Blood Pressure was measured in millimeters of mercury (mmHg) prior to study drug administration and seven days after. The results express the change from baseline (defined as the last measurement prior to the first dose of study drug) to Dose 3.
Time Frame: Change from Baseline to 7 days after study drug administration of Dose 3. Three (3) months
Population: Only participants having received all 3 doses are analyzed and presented.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 4 | 1 | 13 | 7 | 1 | 2
mmHg
  Diastolic | 0.5 (5.74) | 2.0 (0.0) | 2.6 (9.55) | 1.3 (6.47) | 6.0 (0.0) | 6.0 (0.0)
  Systolic | -5.5 (12.61) | 11.0 (0.0) | 5.4 (14.36) | 2.7 (19.81) | 5.0 (0.0) | 2.0 (2.83)

7. Primary Outcome: Assessment of Cellular Immunogenicity Analyses
Description: Assessment of positive CMV IFNγ ELISPOT results for pp65 and gB defined by Spot forming cells / mio PBMC per CMV Management Strategy and Doses Before Transplant
Time Frame: 15 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: SFC/10e6 PBMC
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
SFC/10e6 PBMC
  CMV ELISPOT pp65 (2 Doses): number analyzed (Participants) | 1 | 0 | 3 | 3 | 0 | 0
  CMV ELISPOT pp65 (2 Doses) | 83.0 [83 to 83] |  | 30.7 [15 to 50] | 15.0 [15 to 15] |  |
  CMV ELISPOT pp65 (3 Doses): number analyzed (Participants) | 0 | 0 | 3 | 2 | 1 | 1
  CMV ELISPOT pp65 (3 Doses) |  |  | 95.3 [88 to 105] | 15.0 [15 to 15] | 4145.0 [4145 to 4145] | 3897.0 [3897 to 3897]
  CMV ELISPOT gB (2 Doses): number analyzed (Participants) | 1 | 0 | 2 | 3 | 0 | 0
  CMV ELISPOT gB (2 Doses) | 78.0 [78 to 78] |  | 37.5 [22 to 53] | 11.0 [3 to 15] |  |
  CMV ELISPOT gB (3 Doses): number analyzed (Participants) | 0 | 0 | 4 | 2 | 1 | 1
  CMV ELISPOT gB (3 Doses) |  |  | 59.3 [25 to 112] | 15.0 [15 to 15] | 615.0 [615 to 615] | 1840.0 [1840 to 1840]

8. Secondary Outcome: Time to Clinically Significant CMV Infection.
Description: Measure the time to clinically significant CMV infection, CMV disease, and CMV syndrome. Time to infection was defined as the number of days of the first quantifiable result above the LLOQ monitored for 12 months after transplantation.
Time Frame: 12 months
Population: the number of participants analyzed differs from the total number of participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
days
  CMV Infection: number analyzed (Participants) | 5 | 2 | 6 | 3 | 1 | 2
  CMV Infection | 50.2 (24.05) | 83.0 (69.30) | 256.2 (20.82) | 248.0 (84.59) | 171.0 (0.00) | 15.0 (0.00)
  CMV Syndrome: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 0
  CMV Syndrome | 66.0 (33.94) |  | 277.0 (0.00) |  |  |
  CMV Disease: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 1
  CMV Disease | 62.5 (38.89) |  | 277.0 (0.00) |  | 0 (0) | 0 (0)

9. Secondary Outcome: Number of Participants With CMV Viremia Requiring Anti Viral Therapy
Description: Measure the number of patients with CMV viremia requiring anti viral therapy for CMV seronegative (-) recipients awaiting kidney transplantation from a CMV seropositive (+) donor and to be treated prophylactically for CMV post transplant.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
Participants | 5 | 2 | 5 | 2 | 1 | 1

10. Secondary Outcome: The Time to CMV Viremia Requiring Anti Viral Therapy.
Description: Measure the time to CMV viremia requiring anti viral therapy for CMV seronegative (-) recipients awaiting kidney transplantation from a CMV seropositive (+) donor and to be treated prophylactically for CMV post transplant.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
days | 53.6 (25.13) | 129.0 (124.45) | 259.2 (21.74) | 259.0 (18.38) | 171.0 (0.00) | 15.0 (0.00)

11. Secondary Outcome: Number of Participants Requiring Anti-CMV Therapy
Description: Measure the number of participants requiring anti-CMV therapy (at therapeutic doses) in CMV seropositive (+) recipients awaiting kidney transplant.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
Participants | 5 | 2 | 4 | 2 | 1 | 1

12. Secondary Outcome: The Duration of Anti-CMV Therapy Courses Required.
Description: Measure duration (in days) of anti-CMV therapy courses (at therapeutic doses) required in CMV seropositive (+) recipients awaiting kidney transplant.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 1 | 1
days | 154.2 (77.43) | 89.0 (91.92) | 87.0 (47.17) | 72.0 (24.04) | 198.0 (NA) — No Standard Deviation when one patient analyzed. | 20.0 (NA) — No Standard Deviation when one patient analyzed.

13. Secondary Outcome: Number of Participants With Organ Rejection
Description: Assessment of number of participants with graft failure leading to biopsy-confirmation rejection of organ post transplantation.
Time Frame: Up to 12 months post transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 10 | 4 | 25 | 14 | 6 | 3
Participants | 1 | 0 | 3 | 1 | 0 | 0

14. Secondary Outcome: Time to Organ Rejection
Description: Measurement of time (in days) between transplantation and graft failure leading to biopsy-confirmation rejection of organ
Time Frame: Up to 12 months post transplantation
Population: Number of participants analyzed is based on Secondary Outcome Measure #13. Only participants with organ rejection can be analyzed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
Number analyzed (Participants) | 1 | 0 | 3 | 1 | 0 | 0
days | 59.0 (NA) — Only one participant analyzed. |  | 126.3 (193.81) | 34.0 (NA) — only one participant analyzed. |  |

ADVERSE EVENTS:
Time Frame: Up to 15 months
Arm/Group | HB-101 Vaccine Preemptive | Placebo Preemptive | HB-101 Vaccine Prophylactic | Placebo Prophylactic | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management | HB-101 Vaccine: CMV (+) Patients-Preemptive Management
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 1/34 | 0/17 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/11 | 2/4 | 14/34 | 5/17 | 2/10 | 2/4
Other Adverse Events (participants affected / at risk) | 6/11 | 3/4 | 22/34 | 12/17 | 6/10 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HB-101 Vaccine Preemptive (N=11) | Placebo Preemptive (N=4) | HB-101 Vaccine Prophylactic (N=34) | Placebo Prophylactic (N=17) | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management (N=10) | HB-101 Vaccine: CMV (+) Patients-Preemptive Management (N=4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acute Myocardial Infraction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Agina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
HPT Tertiary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
GI Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Kidney Transplant Rejection (Immune system disorders) | 2 | 0 | 2 | 1 | 0 | 0
Transplant Rejection (Immune system disorders) | 0 | 0 | 2 | 1 | 2 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
CMV Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
CMV Viraemia (Infections and infestations) | 1 | 1 | 1 | 3 | 0 | 0
Enterobacter Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
UTI (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
AKI (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal Artery Thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal Tubular Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
DM Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HB-101 Vaccine Preemptive (N=11) | Placebo Preemptive (N=4) | HB-101 Vaccine Prophylactic (N=34) | Placebo Prophylactic (N=17) | HB-101 Vaccine: CMV (+) Patients-Prophylactic Management (N=10) | HB-101 Vaccine: CMV (+) Patients-Preemptive Management (N=4)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood IgA Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
CMV Test Positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Urine Output Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypomagesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophophataemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
CKD-Mineral and Bone Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 3 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Donor-Specific Antibody Present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Calcium Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Folate Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urethral Spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03629080/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03629080/SAP_001.pdf